CLINICAL TRIAL: NCT00735696
Title: A Phase 2, Open-label Study of IMC-1121B in Combination With Paclitaxel and Carboplatin as First-line Therapy in Patients With Stage IIIB/IV Non-small Cell Lung Cancer
Brief Title: A Study of Ramucirumab (IMC-1121B) With Paclitaxel and Carboplatin in Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13914; 2007-006715-22 (EudraCT Number); CP12-0708 (Other: ImClone Systems); I4T-IE-JVBJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Results first posted 2014-12-29 (Estimated); Last update posted 2014-12-29 (Estimated); Status verified 2014-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; Lung; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Ramucirumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ramucirumab + paclitaxel + carboplatin (Experimental): Participants will receive ramucirumab in combination with paclitaxel and carboplatin until disease progression, the development of an unacceptable toxicity, or other withdrawal criteria, for up to six cycles (3 weeks per cycle).
  In the absence of any withdrawal criteria, participants will continue to receive ramucirumab monotherapy every 3 weeks, provided there is ongoing evidence of benefit upon review every 6 weeks.
  Interventions: Biological: Ramucirumab; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Biological: Ramucirumab — 10 milligrams per kilogram (mg/kg), intravenous (IV) infusion, on Day 1 of each 21-day cycle.
  Other Names: IMC-1121B; LY3009806
Drug: Paclitaxel — 200 milligrams per meter squared (mg/m^2), administered intravenously (IV) following the ramucirumab infusion, on day 1 of each 21-day cycle, for up to six cycles.
Drug: Carboplatin — Administered after paclitaxel, as an intravenous infusion (IV), over 30 minutes on day 1 of each 21-day cycle, for up to six cycles. The dose to be administered is calculated based on the participant's actual body weight at time of treatment and the area under the curve (AUC) dosing. The target AUC for carboplatin treatment is AUC=6.

SUMMARY:
The purpose of this study is to evaluate the progression-free survival (PFS) rate at 6 months of ramucirumab administered in combination with paclitaxel and carboplatin as first-line therapy for Stage IIIB or IV non-small cell lung cancer

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) accounts for 75-80% of all lung cancers. The advanced stages are associated with poor survival rates, a median survival rate of approximately 3.9 months if left untreated.

Angiogenesis is a process for wound healing and restoring blood flow to tissues after injury. It is the physiological process involving the growth of new blood vessels from pre-existing vessels. Angiogenesis may be promoted by growth factors and in diseases such as cancer, where growth factors are over expressed, the body loses the ability to maintain a balanced angiogenesis. This may embellish the existing supplies of blood; potentially increasing the delivery of oxygen and nutrients supplies for cancer growth and survival.

Ramucirumab is an angiogenesis inhibitor; and is believed to block the promotion of the growth factor to form new blood vessels, thus reducing the blood supply to the cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC
* Advanced NSCLC
* Measurable disease (as defined by Response Evaluation Criteria in Solid Tumors [RECIST 1.0])
* Eastern Cooperative Oncology Group (ECOG) Performance Status is ≤ 1
* Age ≥ 18 years
* Adequate hematologic function = an absolute neutrophil count (ANC) ≥ 1500/μL, hemoglobin ≥ 9 g/dL, and a platelet count ≥ 100,000/microliter (μL)
* Adequate hepatic function = a total bilirubin ≤ 1.5 mg/dL transaminases and alkaline phosphatase ≤ 5 x the upper limit of normal (ULN)
* Adequate renal function serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance (CrCl) > 60 mL/minute, and urine dipstick for protein < 1+ (ie, either 0 or trace)
* Adequate coagulation function, INR ≤ 1.5 and a partial thromboplastin time (PTT) ≤ 5 seconds above ULN
* Adequate contraception
* Signed informed consent

Exclusion Criteria:

* Untreated CNS metastases
* Prior bevacizumab therapy
* Radiologically documented evidence of major blood vessel invasion or encasement by cancer
* Prior systemic chemotherapy for Stage IIIB/IV NSCLC
* Prior systemic chemotherapy or radiation therapy for Stage I-IIIA NSCLC < 1 year prior
* Any concurrent malignancy other than basal cell skin cancer, or carcinoma in situ of the cervix
* Concurrent treatment with other anticancer therapy, including other chemotherapy, immunotherapy, hormonal therapy, radiotherapy, chemoembolization, or targeted therapy
* Ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Uncontrolled thrombotic or hemorrhagic disorders
* Poorly-controlled hypertension
* Chronic daily treatment with aspirin (> 325 mg/day) or other known inhibitors of platelet function
* History of gross hemoptysis (defined as bright red blood or ≥ 1/2 teaspoon)
* Serious non-healing wound, ulcer, or bone fracture
* Undergone major surgery or subcutaneous venous access device placement. Post-operative bleeding complications or wound complications from a surgical procedures performed in the last 2 months
* Elective or a planned major surgery to be performed during the course of the trial
* Peripheral neuropathy ≥ Grade 2 (National Cancer Institute Common Toxicity Criteria for Adverse Events, Version 3.0 [NCI-CTCAE v 3.0])
* If female, is pregnant or lactating
* Radiographic evidence of intratumor cavitation
* Grade 3-4 gastrointestinal bleeding within 3 months prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-01; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (9):
- United States (7):
  - ImClone Investigational Site, Beverly Hills, California
  - ImClone Investigational Site, San Francisco, California
  - ImClone Investigational Site, Aurora, Colorado
  - ImClone Investigational Site, New York, New York
  - ImClone Investigational Site, The Bronx, New York
  - ImClone Investigational Site, San Antonio, Texas
  - ImClone Investigational Site, Seattle, Washington
- United Kingdom (2):
  - ImClone Investigational Site, Cambridge
  - ImClone Investigational Site, London

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 52 participants signed informed consent
Groups:
- Ramucirumab + Paclitaxel + Carboplatin: ramucirumab: 10 mg/kg administered intravenously on day 1 of each 21-day cycle.
  paclitaxel: 200 mg/m^2 administered intravenously on day 1 of each 21-day cycle for up to six cycles.
  carboplatin: administered intravenously on day 1 of each 21-day cycle, dose calculated based on the participant's body weight.
  Participants received ramucirumab in combination with paclitaxel and carboplatin until disease progression, the development of an unacceptable toxicity, or other withdrawal criteria, for up to six cycles (3 weeks per cycle). In the absence of any withdrawal criteria, participants continued to receive ramucirumab monotherapy every 3 weeks, provided there was ongoing evidence of benefit upon review every 6 weeks.
Period: Overall Study
Arm/Group | Ramucirumab + Paclitaxel + Carboplatin
Started | 41
Received Any Quantity of Study Drug | 40
Completed | 39
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Enrolled but never Treated | 1

BASELINE CHARACTERISTICS:
Population: Modified intent to treat population (mITT): All participants who received any quantity of study drug.
Groups:
- Ramucirumab + Paclitaxel + Carboplatin: ramucirumab: 10 mg/kg administered intravenously on day 1 of each 21-day cycle.
  paclitaxel: 200 mg/m^2 administered intravenously on day 1 of each 21-day cycle for up to six cycles.
  carboplatin: administered intravenously on day 1 of each 21-day cycle, dose calculated based on the participant's body weight.
  Participants will receive ramucirumab in combination with paclitaxel and carboplatin until disease progression, the development of an unacceptable toxicity, or other withdrawal criteria, for up to six cycles (3 weeks per cycle). In the absence of any withdrawal criteria, participants will continue to receive ramucirumab monotherapy every 3 weeks, provided there is ongoing evidence of benefit upon review every 6 weeks.
Arm/Group | Ramucirumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 34
  Black or African American | 4
  Asian | 2
Region of Enrollment [Number; unit: participants]
  United States | 36
  United Kingdom | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Are Progression-free (PFS) at 6 Months
Description: Data presented are the percentage of participants without disease progression or death at 6 months. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0). Progressive disease was defined as having at least a 20% increase in sum of longest diameter of target lesions or the appearance of one or more new lesions and/or unequivocal progression of existing nontarget lesions.
Time Frame: 6 months
Population: Modified intent to treat population (mITT): All participants who received any quantity of study drug.
  Nine participants were censored.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ramucirumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 40
percentage of participants | 59.0 [41.3 to 72.9]

2. Secondary Outcome: Summary of Participants Reporting Adverse Events
Description: Data presented are the number of participants who experienced ramucirumab related treatment-emergent adverse events (TEAE), treatment related serious adverse events (SAE), or any Grade 3 or higher TEAE; any TEAE leading to discontinuation of ramucirumab treatment, and any TEAE leading to dose modification ramucirumab. A summary of SAEs and other nonserious AEs, regardless of causality, is located in the Reported Adverse Event section.
Time Frame: Baseline up to 32.5 months
Population: Safety Population: All participants who received any quantity of study drug.
Measure: Number; unit: participants
Arm/Group | Ramucirumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 40
participants
  Any ramucirumab related TEAE | 34
  Any ramucirumab related Serious TEAE | 8
  Any ramucirumab related Grade >= 3 TEAE | 15
  Any TEAE Leading to Discontinuation of ramucirumab | 13
  TEAE Leading to Dose Modification of ramucirumab | 24
  Any ramucirumab related TEAE with Outcome of Death | 0

3. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) (Objective Response Rate ([ORR])
Description: Objective response is Complete Response (CR) + Partial Response (PR), as classified by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST 1.0) guidelines. CR is a disappearance of all target and non-target lesions; PR is at least a 30% decrease in the sum of the longest diameter of target lesions without new lesions and progression of non-target lesions. Objective response rate is calculated as a total number of participants with CR or PR divided by the total number of participants with measurable disease, multiplied by 100.
Time Frame: First dose to measured progressive disease or death due to any cause up to 32.5 months
Population: Modified intent to treat population (mITT): All participants who received any quantity of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ramucirumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 40
percentage of participants | 55.0 [38.5 to 70.7]

4. Secondary Outcome: Duration of Response
Description: The duration of a complete response (CR) or partial response (PR) was defined as the time from first objective status assessment of CR or PR to the first time of progression, initiation of additional antitumor therapy is first reported, or death as a result of any cause. CR was defined as the disappearance of all target lesions. PR was defined as having at least a 30% decrease in sum of longest diameter of target lesions.
Time Frame: First dose up to 32.5 months
Population: Participants who had tumor response. Two participants who had tumor response did not progress by the data cut-off date, therefore were censored for duration of response analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 22
months | 5.54 [4.27 to 8.21]

5. Secondary Outcome: Overall Survival (OS) at 1 Year
Description: Data presented are the percentage of participants surviving at least 12 months after first dose of study medication.
Time Frame: First dose to 1 year
Population: Modified intent to treat population (mITT): All participants who received any quantity of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ramucirumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 40
percentage of participants | 74.6 [57.9 to 85.4]

6. Secondary Outcome: Progression-free Survival (PFS)
Description: Defined as the time from date of first dose of study medication to the first documented disease progression as defined by Response Evaluation Criteria In Solid Tumors (RECIST 1.0), initiation of additional antitumor therapy was first reported or death due to any cause.
  Participants who did not progress, who discontinued treatment for toxicity or a reason other than documented progression, or who were lost to follow-up before documented progression or death were censored at date of last tumor assessment. Participants who started new therapeutic anticancer treatment prior to documented progression or death were censored at date of last tumor assessment prior to new therapeutic anticancer therapy.
Time Frame: First dose to measured progressive disease or death due to any cause, up to 32.5 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 40
months | 7.85 [5.49 to 9.86]

7. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the first dose of study medication to the date of death from any cause. Participants who were alive at the end of the follow-up period or lost to follow-up were censored on the last date the patient was known to be alive.
Time Frame: First dose to death due to any cause, up to 32.5 months
Population: Modified intent to treat population (mITT): All participants who received any quantity of study drug.
  Fourteen participants were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 40
months | 16.85 [14.82 to 28.58]

8. Secondary Outcome: Serum Anti-Ramucirumab Antibody Assessment
Description: The number of participants who developed treatment emergent antibody responses to ramucirumab after baseline.
Time Frame: Week 15 (Cycle 5)
Population: Participants who had Anti-Ramucirumab Antibody assessment at week 15 (cycle 5).
Measure: Number; unit: participants
Arm/Group | Ramucirumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 29
participants | 1

9. Secondary Outcome: Maximum Concentration of Ramucirumab (Cmax)
Time Frame: Week 18 (Cycle 6), at 1-Hour Post End of Infusion
Population: Participants who received any quantity of study medication and had evaluable concentration data at the specified time point.
Measure: Mean (Standard Deviation); unit: micrograms/milliliter (mcg/mL)
Arm/Group | Ramucirumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 8
micrograms/milliliter (mcg/mL) | 372 (82.9)

ADVERSE EVENTS:
Arm/Group | Ramucirumab + Paclitaxel + Carboplatin
Serious Adverse Events (participants affected / at risk) | 19/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab + Paclitaxel + Carboplatin (N=40)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 4 (5)
NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
CHILLS (General disorders) | 1 (1)
FATIGUE (General disorders) | 1 (1)
INFUSION RELATED REACTION (General disorders) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1)
ANAPHYLACTIC REACTION (Immune system disorders) | 1 (1)
CATHETER SEPSIS (Infections and infestations) | 2 (2)
EMPYEMA (Infections and infestations) | 1 (1)
PERIANAL ABSCESS (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1)
SINUSITIS (Infections and infestations) | 1 (1)
CONVULSION (Nervous system disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1)
SYNCOPE VASOVAGAL (Nervous system disorders) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab + Paclitaxel + Carboplatin (N=40)
ANAEMIA (Blood and lymphatic system disorders) | 5 (6)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2)
LEUKOPENIA (Blood and lymphatic system disorders) | 3 (4)
NEUTROPENIA (Blood and lymphatic system disorders) | 13 (28)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 13 (42)
TACHYCARDIA (Cardiac disorders) | 2 (3)
VISION BLURRED (Eye disorders) | 2 (2)
VISUAL ACUITY REDUCED (Eye disorders) | 2 (2)
CONSTIPATION (Gastrointestinal disorders) | 16 (24)
DIARRHOEA (Gastrointestinal disorders) | 14 (19)
DRY MOUTH (Gastrointestinal disorders) | 2 (2)
DYSPEPSIA (Gastrointestinal disorders) | 3 (4)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 6 (6)
GINGIVAL PAIN (Gastrointestinal disorders) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 23 (38)
STOMATITIS (Gastrointestinal disorders) | 6 (6)
VOMITING (Gastrointestinal disorders) | 14 (14)
ASTHENIA (General disorders) | 2 (4)
CHILLS (General disorders) | 2 (2)
FATIGUE (General disorders) | 29 (58)
INFLUENZA LIKE ILLNESS (General disorders) | 2 (3)
INFUSION RELATED REACTION (General disorders) | 7 (10)
MUCOSAL INFLAMMATION (General disorders) | 2 (2)
NON-CARDIAC CHEST PAIN (General disorders) | 9 (9)
OEDEMA PERIPHERAL (General disorders) | 11 (12)
PAIN (General disorders) | 2 (2)
PYREXIA (General disorders) | 4 (6)
TEMPERATURE INTOLERANCE (General disorders) | 2 (5)
CELLULITIS (Infections and infestations) | 3 (3)
FOLLICULITIS (Infections and infestations) | 3 (5)
NASOPHARYNGITIS (Infections and infestations) | 2 (3)
PNEUMONIA (Infections and infestations) | 2 (2)
TOOTH ABSCESS (Infections and infestations) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3)
URINARY TRACT INFECTION (Infections and infestations) | 4 (4)
WEIGHT DECREASED (Investigations) | 7 (10)
ANOREXIA (Metabolism and nutrition disorders) | 10 (12)
DEHYDRATION (Metabolism and nutrition disorders) | 5 (6)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 5 (5)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 2 (2)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 16 (21)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (4)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 3 (3)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 (2)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 3 (4)
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 2 (2)
MYALGIA (Musculoskeletal and connective tissue disorders) | 11 (15)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 (9)
BALANCE DISORDER (Nervous system disorders) | 2 (2)
DIZZINESS (Nervous system disorders) | 5 (6)
DYSGEUSIA (Nervous system disorders) | 6 (6)
HEADACHE (Nervous system disorders) | 11 (14)
HYPOAESTHESIA (Nervous system disorders) | 3 (5)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 27 (44)
SYNCOPE (Nervous system disorders) | 2 (2)
ANXIETY (Psychiatric disorders) | 7 (7)
DEPRESSION (Psychiatric disorders) | 5 (6)
INSOMNIA (Psychiatric disorders) | 4 (4)
PROTEINURIA (Renal and urinary disorders) | 4 (10)
PELVIC DISCOMFORT (Reproductive system and breast disorders) | 2 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 10 (13)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 4 (4)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 9 (9)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 5 (5)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 12 (15)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 3 (3)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2 (3)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3 (3)
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 2 (2)
ORTHOPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 (4)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 4 (4)
ALOPECIA (Skin and subcutaneous tissue disorders) | 23 (37)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 3 (3)
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 (2)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 6 (6)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 2 (2)
NAIL DISCOLOURATION (Skin and subcutaneous tissue disorders) | 2 (2)
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 2 (2)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2)
RASH (Skin and subcutaneous tissue disorders) | 8 (8)
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 2 (2)
SKIN LESION (Skin and subcutaneous tissue disorders) | 3 (3)
URTICARIA (Skin and subcutaneous tissue disorders) | 2 (2)
HYPERTENSION (Vascular disorders) | 6 (6)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 2 (2)
PHLEBITIS (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.